CLINICAL TRIAL: NCT03990220
Title: A Nutritional Trial on Effect of Probiotic Yoghurt Containing Lactobacillus Rhamnosus Yoba 2012 on Respiratory Tract Infection and Other Health Outcomes Among Children Aged 3-6 Years in Southwest Uganda
Brief Title: A Nutritional Trial on Effect of L. Rhamnosus Yoba on RTI and Other Health Outcomes Among Children (3-6 Years) in Uganda
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: VU University of Amsterdam (Other)
Collaborators: Yoba for Life Foundation (Unknown)
Responsible Party: Principal Investigator, Remco Kort, Professor, VU University of Amsterdam
Other Study IDs: 01/09-18
Record Dates: First submitted 2019-05-12; First posted 2019-06-18 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-11

CONDITIONS: Skin Diseases; Respiratory Tract Infections; Diarrhea
Keywords: probiotics; Lactobacillus rhamnosus yoba 2012; Skin diseases; Respiratory Tract Infections; School absenteeism; Diarrhea; Anthropometric indicators
MeSH Terms: conditions — Skin Diseases; Respiratory Tract Infections; Diarrhea

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Biospecimen Retention: None Retained — Urine Samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment: 500 children, 3-6 years old attending pre-primary school in Southwest Uganda, who recently decided to start the consumption of yoghurt containing Lactobacillus rhamnosus, 100 ml per day, on any school day (i.e. monday - friday with the exception of school holidays).
  Interventions: Dietary Supplement: Lactobacillus rhamnosus yoba 2012
- Control: 500 children, 3-6 years old attending pre-primary school in Southwest Uganda, who recently decided to start the consumption of milk, 100 ml per day, on any school day (i.e. monday - friday with the exception of school holidays).

INTERVENTIONS:
Dietary Supplement: Lactobacillus rhamnosus yoba 2012 — Probiotics are defined by the Food and Agricultural Organization (FAO)/WHO as "live microorganisms, which when consumed in adequate amounts, confer a health benefit on the host". Lactobacillus rhamnosus GG (LGG) is the most documented probiotic bacteria, with many proven unique characteristics and therewith associated health benefits. No adverse effects of the consumption of LGG in healthy infants have been reported. The Lactobacillus rhamnosus yoba containing yoghurt drink, which is locally produced and subsequently consumed by resource-poor communities in rural Uganda has been described. The strain used in this intervention is a generic variant of LGG, called Lactobacillus rhamnosus yoba 2012. LGG is consumed as part of food all over the world, and is not a drug.
  Other Names: Lactobacillus rhamnosus GG
  Groups: Treatment

SUMMARY:
This is a nutritional observational trial with two arms: 1) Intervention arm of Probiotic Yoghurt containing Lactobacillus rhamnosus yoba 2012 and 2) Control arm of milk. About 500 children in each arm will be enrolled. Children will be enrolled in the yoghurt or the milk arm, based on the preference of the school and the parents in response to a sensitization campaign of a non-governmental organization (NGO) in the region. This selection will therefore be non-randomized and non-blinded. Within one school, all children will be enrolled in the same arm. The children will be monitored for 3 weeks in the baseline. Subsequently, the children will consume either 100ml of yoghurt or 100ml of milk, once per day for five days per week for nine weeks, while being continuously monitored. The milk and the yoghurt will be locally sourced in the district where the schools are located.

DETAILED DESCRIPTION:
This is an observational nutritional trial with two arms: 1) Intervention arm of Probiotic Yoghurt containing Lactobacillus rhamnosus yoba 2012 and 2) Control arm of milk. About 500 children in each arm will be enrolled. Children will be enrolled in the yoghurt or the milk arm, based on the preference of the school and the parents in response to a sensitization campaign of an NGO in the region. This selection will therefore be non-randomized and non-blinded. Within one school, all children will be enrolled in the same arm. The children will be monitored for 3 weeks in the baseline. Subsequently, the children will consume either 100ml of yoghurt or 100ml of milk, once per day for five days per week for nine weeks, while being continuously monitored. The milk and the yoghurt will be locally sourced in the district where the schools are located. Monitoring and data collection tools include:

1. Baseline, midline and end line questionnaire administered to parents to identify confounding factors (e.g. use of medication and diet from home) of treatment and control group.
2. Weight, height, mid-upper-arm circumference MUAC and head circumference measurements every 4 weeks for 3 months in both the treatment and control groups (total 4 times). One point measurement will be taken 6 months after the study.
3. Daily monitoring of the incidence of RTIs, diarrhoea, skin rashes or other diseases in treatment and control groups by teachers with confirmation of a nurse in a mobile app.

Children from pre-primary institutions in which both the management and the parents have recently decided to purchase either milk or yoghurt for the pupils on regular basis will be recruited. The study subjects (children) are recruited at these institutions. Only children from parents who have agreed to contribute to the consumption of milk / yoghurt and who have furthermore consented for their children to be measured and monitored for the purpose of the current study will be recruited. The parent is free to provide his/her child with milk / yoghurt, even if the parent does not consent for the child to take part in the study.

The study will start three weeks before either milk or yoghurt consumption commences, in order to establish a solid baseline. With the help of tablets and a specially designed app, nurses will keep track of their pupils' health by tracking incidence of diarrhoea, respiratory tract infections, skin rashes and other diseases. Teachers will keep track of the daily attendance of pupils.

Measurements of weight, height, MUAC and head circumference will be measured by a nurse every four weeks, starting three weeks prior to the start of the consumption of either milk or yoghurt. The measurements will be conducted with the help of Standard Operations Procedures as provided by Life Study and analysed with the help of World Health Organization (WHO) guidelines.

During these 3 months in which the children will be monitored, a questionnaire will be administered to the parents of the children at the start, middle and end of the study. The primary objective and content of the questionnaire is related to diet of the children outside school, in order to determine whether there are significant differences between the diets of the children in the treatment group and in the control group. The questionnaires will furthermore include questions about absenteeism and causes thereof, incidence of diarrhoea, Respiratory Tract Infections or any other diseases, and the use of any type of drug or treatment, in order to verify and supplement the information provided by the class-teacher.

ELIGIBILITY:
Inclusion Criteria:

* During interactions with the pre-primary institutions prior to the study, the parents of the children have agreed to pay for their child to either take milk or probiotic yoghurt (100ml five times per week).
* Parents are willing to provide written consent for their child to participate in the study, and children are willing to provide assent

Exclusion Criteria:

* The child does not comply with the inclusion criteria
* The child has an aversion against yoghurt or milk
* The child is lactose-intolerant as indicated by the parent, or has any other medical condition that will prevent him/her from taking yoghurt or milk.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children 3-6 years old attending pre-primary schools in the districts Kiruhura, Lyantonde, Sheema, Bushenyi, Mbarara, Isingiro or Ntungamo in Southwest Uganda. Children of all genders and all health statuses are enrolled.
Sampling Method: Non-Probability Sample
Enrollment: 1116 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-09-15 (Actual); Study Completion 2020-06-01 (Estimated)

PRIMARY OUTCOMES:
The number of children on each individual day that suffers from Respiratory Tract Infections | 3 months
  To compare the incidence of respiratory tract infections among children aged 3-6 years in Southwest Uganda before, during and after an intervention with probiotic yoghurt containing Lactobacillus rhamnosus yoba

SECONDARY OUTCOMES:
Changes in weight of children during the study period | 3 months
  To monitor changes in weight of children aged 3-6 years in Southwest Uganda who consume yoghurt containing Lactobacillus rhamnosus yoba.
Changes in height of the children during the study period | 3 months
  To monitor changes in height of children aged 3-6 years in Southwest Uganda who consume yoghurt containing Lactobacillus rhamnosus yoba.
The number of children on each individual day that suffers from Diarrhea | 3 months
  To compare the incidence of diarrhea among the children before, during and after the intervention.
The number of children on each individual day that suffers from any form of skin diseases | 3 months
  To compare the incidence of skin diseases among the children before, during and after the intervention.
The number of children on each individual day that is Absent | 3 months
  To compare absenteeism as a result of sickness among the children before, during and after the intervention.

CONTACTS AND LOCATIONS:
Overall Officials: Remco Kort, PhD, Principal Investigator — VU Amsterdam
Locations (10):
- Uganda (10):
  - BDA Nursery and Primary School, Ishaka, Bushenyi
  - Jireh Junior School, Ishaka, Bushenyi
  - Itojo Nusery and Primary School, Itojo, Ntungamo
  - Queen and King Nursery and Primary School, Itojo, Ntungamo
  - Blue Sight Primary School, Kabwohe, Sheema
  - Faith Memorial Nursery and Primary School, Bushenyi
  - Hanny Nusery and Primary School, Isingiro
  - St. Eliza Excell Nursery and Primary School, Isingiro
  - St. Francis Nursery and Primary School, Lyantonde
  - Mbarara Progressive Nursery and Primary School, Mbarara

IPD SHARING:
Plan to Share IPD: No
Data will be uploaded to the online respiratory of the app as developed by Omnitech. This data will only be accessible to the researchers who have been granted the password. Besides, data will be primarily entered in excel, and analysed with the help of Statistical Package for Social Sciences (SPSS). Data will be cross validated by the different researchers involved. Data will be handled confidentially and anonymously, provided with a code and will be only accessible to the researchers.
  The data collection app will create monthly health reports, which will be shared with parents to enable them to closely monitor the health and development of their children.

REFERENCES:
- [Background] Dezateux, C., Williams, J., Walton, S., Wells, J., 2016. Life Study Standard Operating Procedures: Adult Anthropometry.
- [Background] Williams, J., Walton, S., Wells, J., 2016. Life Study Standard Operating Procedures: Infant Anthropometry.
- [Background] World Health Organization (Ed.), 2007. WHO child growth standards: head circumference-for-age, arm circumference-for-age, triceps skinfold-for-age and subscapular skinfold-for-age: methods and development. World Health Organization, Geneva
- [Background] World Health Organization (Ed.), 2006. WHO child growth standards: length/height-for-age, weight-for-age, weight-for-length, weight-for-height and body mass index-for-age ; methods and development. WHO Press, Geneva.
- [Background] Pineiro M, Stanton C. Probiotic bacteria: legislative framework-- requirements to evidence basis. J Nutr. 2007 Mar;137(3 Suppl 2):850S-3S. doi: 10.1093/jn/137.3.850S. PMID 17311986
- [Background] Petschow BW, Figueroa R, Harris CL, Beck LB, Ziegler E, Goldin B. Effects of feeding an infant formula containing Lactobacillus GG on the colonization of the intestine: a dose-response study in healthy infants. J Clin Gastroenterol. 2005 Oct;39(9):786-90. doi: 10.1097/01.mcg.0000177245.53753.86. PMID 16145341
- [Background] Scalabrin D, Harris C, Johnston WH, Berseth CL. Long-term safety assessment in children who received hydrolyzed protein formulas with Lactobacillus rhamnosus GG: a 5-year follow-up. Eur J Pediatr. 2017 Feb;176(2):217-224. doi: 10.1007/s00431-016-2825-4. Epub 2016 Dec 15. PMID 27975116
- [Background] Kort R, Westerik N, Mariela Serrano L, Douillard FP, Gottstein W, Mukisa IM, Tuijn CJ, Basten L, Hafkamp B, Meijer WC, Teusink B, de Vos WM, Reid G, Sybesma W. A novel consortium of Lactobacillus rhamnosus and Streptococcus thermophilus for increased access to functional fermented foods. Microb Cell Fact. 2015 Dec 8;14:195. doi: 10.1186/s12934-015-0370-x. PMID 26643044
- [Background] Kort R, Sybesma W. Probiotics for every body. Trends Biotechnol. 2012 Dec;30(12):613-5. doi: 10.1016/j.tibtech.2012.09.002. Epub 2012 Sep 29. No abstract available. PMID 23031355